CLINICAL TRIAL: NCT00789763
Title: Open-label, Multicentric Phase I-II Trial to Evaluate the Efficacy and Safety of the Combination of Sorafenib (BAY 43-9006), Gemcitabine and Concurrent Radiotherapy, in Locally Advanced Pancreatic Carcinoma
Brief Title: Phase I-II to Evaluate Efficacy/Safety of Sorafenib+Gemcitabine+Radiotherapy in Locally Advanced Pancreatic Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Grupo Espanol Multidisciplinario del Cancer Digestivo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEMCAD 0701
Record Dates: First submitted 2008-11-11; First posted 2008-11-13 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; Pancreatic cancer locally advanced
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Radiotherapy; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sorafenib + gemcitabine + radiotherapy (Experimental)
  Interventions: Drug: Gemcitabine; Radiation: Radiotherapy; Drug: Sorafenib

INTERVENTIONS:
Drug: Gemcitabine — 300 mg/m2/one per week, i.v., during 5 weeks.
Radiation: Radiotherapy — 1.8 Gy/day 5 days per week during 5 weeks (total dose 45Gy)
Drug: Sorafenib — 200-800 mg/day p.o. during 5 weeks
  Other Names: Brand name: nexavar

SUMMARY:
Phase I: Safety profile and to determine maximum tolerated dose (MTD) / Recommended Dose (DR) of Sorafenib in combination with Gemcitabine and Radiotherapy

Phase II: Activity profile evaluating Progression-free rates (PFR) at 6 months, Response rate, Overall survival, Toxicity profile

DETAILED DESCRIPTION:
Safety profile and to determine maximum tolerated dose (MTD) / Recommended Dose (DR) of Sorafenib in combination with Gemcitabine and Radiotherapy

Definition of maximum tolerated dose (MTD):

The MTD is defined as the highest dose level which can be given to 6 patients such that no more than 1 patient experiences a DLT .

Definition of Recommended Dose (DR):

Is the MTD

Definition of Dose-limiting toxicity (DLT):

DLT will be defined as any of the following occurring during the period of treatment and regarded as related to the combination regimen.

* Grade 4 thrombocytopenia persisting greater than 4 days, or with bleeding requiring platelet transfusion
* Grade 4 neutropenia lasting more than 7 days
* Febrile neutropenia (≥ 38.5oC) with an absolute neutrophil count ≤ 1000/mm3
* Any grade 3 or 4 non-hematologic toxicity related to the combination [occurring despite optimal supportive care, if applicable] except hyperglycemia, hypoglycemia, deep venous thrombosis, or hyperbilirubinemia secondary to stent malfunction.
* Hypertension that is symptomatic and not managed by maximal use of three different classes of antihypertensives, or any episode of malignancy hypertension

(Detailed Dose Modifications and G-CSF use in case of febrile neutropenia will be outlined in the full protocol version)

Phase II

Primary objective:

Activity profile evaluating Progression-free rates (PFR) at 6 months

Secondary objective:

Response rate Overall survival Toxicity profile

ELIGIBILITY:
Inclusion Criteria:

1. -Patients with histological or cytological confirmed locally advanced pancreatic adenocarcinoma pancreatic carcinoma or metastatic pancreatic carcinoma for phase I.
2. -Patients with measurable (according to RECIST) disease.
3. -Male or female patients > or = 18 years old
4. -ECOG 0-1
5. -Adequate bone marrow, liver , and renal function: Absolute neutrophil count ( ANC) >= 1,500/mm3 Platelets> or = 100,000/µl Hemoglobin >=9.0 g/dl Total bilirubin < 1.5 x the upper limit of normal. ALT and AST <= 2.5 x upper limit of normal ( <= 5X upper limit of normal for patients with liver involvement ) Serum creatinine <= 1.5 times x the upper limit of normal. Patients with creatinine clearance >= 45mL/min PT( prothrombin time ) or INR( international normalized ratio ) and PTT ( partial thromboplastin time ) < =1.5 x
6. -Women of childbearing potential and men must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation. Men should use adequate birth control for at least six months after the last administration of sorafenib
7. -Signed informed consent prior to any study specific procedures

Exclusion Criteria:

1. -Patients with previous treatment for pancreatic carcinoma
2. -PTV ( planning target volume ) >500 cm3 or 5 cm (maximum diameter)
3. -Patients with known or suspected allergy to iodated contrasts or renal impairment which prevents from radiological tests.
4. -Pregnant or nursing patients. Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment
5. -General medical or psychological conditions that would preclude appropriate informed consent or compliance with the protocol.
6. -Previous cancer that is distinct in primary site or histology from NSCLC except cervical cancer in-situ, treated basal cell carcinoma, superficial bladder tumors (Ta and Tis) or any cancer curatively treated > 3 years prior to study entry
7. -Concurrent treatment with other experimental drugs (within 30 days prior to study entry).
8. -Concurrent treatment with other anti-cancer therapy.
9. -Therapeutic anticoagulation with Vitamin K antagonists such as warfarin or with heparins or heparinoids. Low dose warfarin is permitted if INR is <1.5 . Low dose aspirin is permitted .
10. -Patients with any medical condition which could jeopardize their safety while his participation in the study .
11. -Significant weight loss (> or equal 10% body weight during preceding 6 weeks)
12. -Major surgery within 3 previous weeks, or laparoscopic biopsy or significant traumatic injury within 2 weeks of prior to first dose of study drug.
13. -Known or suspected allergy to sorafenib or any agent given in the course of this trial .
14. -Patients with evidence or history of bleeding diathesis or coagulopathy
15. -Thrombotic or embolic events such as cerebrovascular accident including transient ischemic attacks within the past 6 months
16. -Uncontrolled hypertension defined as systolic blood pressure > 150 mm Hg or diastolic pressure > 90 mm Hg, despite optimal medical management
17. -Cardiac disease: Congestive heart failure > class II NYHA. Patients must not have unstable angina or new-onset angina (began within the last 3 months) or myocardial infarction within the last 6 months
18. -Patients with Child-Pugh class C hepatic impairment
19. -Patients with severe renal impairment (calculated creatinine clearance of < 30 ml/min) or who require dialysis
20. -Active clinically serious infections > CTCAE Grade 2
21. -Serious, non-healing wound, ulcer, or bone fracture
22. -Patients with concomitant ketoconazole, itraconazole,ritonavir,rifampicin or St. John's Wort (Hypericum perforatum).
23. -Known brain metastasis. Patients with neurological symptoms should undergo a CT scan/MRI of the brain to exclude brain metastasis
24. -Any instable condition that may interfere with the patients participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-12; Primary Completion 2011-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
SAFETY | End of Study
EFFICACY | End of Study
TO DETERMINE MTD | Treatment (5 weeks)

SECONDARY OUTCOMES:
RESPONSE (ACCORDING TO RECIST) | End of Study

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Hospital de La Santa Creu I Sant Pau, Barcelona, Barcelona
  - Hospital Clinic I Provincial, Barcelona, Barcelona
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Universitario La Fe, Valencia, Valencia

REFERENCES:
- [Derived] Aparicio J, Garcia-Mora C, Martin M, Petriz ML, Feliu J, Sanchez-Santos ME, Ayuso JR, Fuster D, Conill C, Maurel J. A phase I, dose-finding study of sorafenib in combination with gemcitabine and radiation therapy in patients with unresectable pancreatic adenocarcinoma: a Grupo Espanol Multidisciplinario en Cancer Digestivo (GEMCAD) study. PLoS One. 2014 Jan 9;9(1):e82209. doi: 10.1371/journal.pone.0082209. eCollection 2014. PMID 24416138